CLINICAL TRIAL: NCT02864329
Title: Small RNA Pathways in Mammalian Gametogenesis
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Cornell University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1209013034; 5P50HD076210 (NIH)
Record Dates: First submitted 2016-04-26; First posted 2016-08-12 (Estimated); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Male Infertility
Keywords: Male Infertility; micro RNAs; small interfering RNAs; miRNA; siRNA
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Testicular tissue, penile tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
Basic and clinical research is revealing that various noncoding and small RNAs play important and diverse roles in germ cell development and quality, including X/Y silencing during meiosis, gene regulation, DNA damage responses, and protection of the genome against transposable elements. Indeed, mammalian germ cells are known to harbor multiple small RNA species, including small interfering RNAs (siRNA), microRNAs (miRNA), and germline- specific PIWI- interacting RNAs (piRNA). However, their mechanistic roles in gametogenesis and human infertility are largely uncharacterized. The goal of this study is to elucidate the role of small RNA pathways in the events that give rise to viable euploid gametes. Four projects and three cores are included in this study.

DETAILED DESCRIPTION:
Project 2 (PI: Dr. Darius Paduch): Role of Small RNAs in male infertility. The leading hypothesis of this project is based on extensive preliminary results obtained by this group showing that 70% of miRNA expressed from human testis are highly conserved in humans and rodents. The investigators hypothesize that differentially expressed miRNAs in men with infertility lead to changes in levels of target messenger RNAs (mRNAs) involved in key regulatory pathways in cell biology. The results of this project will lead to better understanding of miRNAs' role in male reproduction and have strong potential to enable the development of new miRNA-based or miRNA-regulating therapies. This project will help to develop new transgenic animals to study miRNA in vivo with implications not only for infertility, but also biology of testicular cancer. Derived RNA based therapies have the potential to be less invasive, less toxic, and more effective in treating these serious and increasingly prevalent conditions.

Core A (PI: Dr. Paula E. Cohen): Administration Core. The main objective of the Administrative Core (Core A) is to provide a structure and support mechanism to the entire Center for Reproductive Genomics (CRG). The Admin core will facilitate interactions across the Ithaca and Manhattan campuses of Cornell University, will encourage research in small RNA biology, both in reproductive medicine and across clinical disciplines, and will promote strong training in reproductive medicine that encourages a translational focus. In general, the Admin core will focus efforts on three major philosophies: translational and innovative research, teaching, and outreach.

Core B (PI: Dr. Andrew Grimson): RNA Sequencing Core. The main objective of the RNA Sequencing Core (RSC) is to provide users with efficient and high quality access to cutting-edge sequencing technologies. These sequencing technologies will be used by all members of this P50-proposal, and made available to other P50-centers. Importantly, all members of this P50 are relying on access to these technologies to achieve their project goals. By centralizing sequencing at the RSC, sequencing will be performed at a lower cost and with greater efficiency that would be possible for individual users.

Core C (PI: Dr. Peter Schlegel): Outreach Core The goals of this outreach core are two-fold: (1) to provide a scientific and technical resource for clinicians interested in embarking on research involving small RNA biology in their physiological system of interest, and (2) to provide outreach to the community by means of a state- of-the-art lecture series. The Innovation Seminars in Reproductive Technologies Series (InSeRT), in order to educate patients about the latest advances in our understanding of the genetic and epigenetic basis for human disease.

ELIGIBILITY:
Inclusion Criteria:

* Men between the ages of 18-90 who have testicular cancer and underwent surgery at Weill Cornell Medicine.

Exclusion Criteria:

* Women, men outside of the age parameters

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men between the age of 18 and 90 who have testicular cancer and underwent surgery for removal at Weill Cornell Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2014-04; Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Using RNA from men with normal spermatogenesis and men with infertility for multiplexed deep sequencing to identify differentially expressed miRNAs | 5 years
  Detect target mRNAs through correlation analysis of actual mRNA expression profiles obtained from the same patients. At the end of the proposed funding period, project 2 will have identified and confirmed a set of approximately 20-30 miRNA:mRNA interactions in male infertility.

CONTACTS AND LOCATIONS:
Overall Officials: Peter N Schlegel, M.D., Principal Investigator — Weill Medical College of Cornell University; Paula E. Cohen, Ph.D., Principal Investigator — Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No